CLINICAL TRIAL: NCT00595790
Title: Phase 3 Study to Compare a Rapid Immunization Regime With the Standard Regime of IC51 as Vaccine for Japanese Encephalitis
Brief Title: Rapid Immunization Study of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IC51-304
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- IC51 2 x 6 mcg (Active Comparator): 2 x 6 mcg (microgram)
  Interventions: Biological: IC51
- IC51 1 x 12 mcg (Active Comparator): 1 x 12 mcg (microgram)
  Interventions: Biological: IC51
- IC51 1 x 6 mcg (Active Comparator): 1 x 6 mcg (microgram)
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51
  Other Names: Japanese Encephalitis purified inactivated vaccine

SUMMARY:
The study investigates a rapid immunization regime of the Japanese Encephalitis vaccine IC51 (JE-PIV) in healthy subjects aged > or = 18 years

DETAILED DESCRIPTION:
This is a multicenter, observer blinded, controlled, randomized phase 3 study. The study population consists of healthy male and female volunteers, aged at least 18 years.

Approximately 375 volunteers will be enrolled at approximately 2 to 3 sites.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent obtained prior to study entry

Exclusion Criteria:

* History of clinical manifestation of any flavivirus infection
* History of vaccination against Japanese encephalitis (JE), Yellow fever and Dengue fever (an anti-JEV neutralizing antibody titer >= 1:10 at baseline is acceptable for inclusion, these subjects will be part of the safety population, but will not be analyzed for immunogenicity in the per-protocol analysis)
* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period or within 30 days preceding the first dose of study vaccine
* Immunodeficiency including post-organ-transplantation or immunosuppressive therapy
* A family history of congenital or hereditary immunodeficiency
* History of autoimmune disease
* Any acute infections within 4 weeks prior to enrollment
* Infection with HIV, Hepatitis B or Hepatitis C
* Pregnancy, lactation or unreliable contraception in female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eder, Mag., Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IC51 2 x 6 mcg | IC51 1 x 12 mcg | IC51 1 x 6 mcg
Started | 125 | 124 (124 subjects randomized to this group, 125 subjects received 1x12 mcg.(Safety Population: N=125)) | 125 (125 subjects randomized to this group, 124 subjects received 1x6 mcg.(Safety Population: N=124))
Completed | 123 (The Participant Flow shows all study participants randomized.Prim. Outcome is based on PP Population) | 123 (The Participant Flow shows all study participants randomized.Prim. Outcome is based on PP Population) | 122 (The Participant Flow shows all study participants randomized.Prim. Outcome is based on PP Population)
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 2 x 6 mcg | IC51 1 x 12 mcg | IC51 1 x 6 mcg | Total
Number analyzed (Participants) | 125 | 125 | 124 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (14.2) | 41.2 (15.0) | 41.6 (14.8) | 40.8 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristics are based on Safety Population: all randomized subjects who received at least one vaccination, analysed using the treatment actually received.
  Participants
    Female | 71 | 65 | 61 | 197
    Male | 54 | 60 | 63 | 177
Region of Enrollment [Number; unit: participants]
  United Kingdom | 58 | 58 | 57 | 173
  Germany | 67 | 67 | 67 | 201

OUTCOME MEASURES:

1. Primary Outcome: SCR (Seroconversion Rate) at Day 56
Description: Seroconversion rate: percentage of subjects with >= 1:10 anti-JEV neutralizing antibody titer
Time Frame: day 56
Population: The Participant Flow shows all study participants randomized. The Primary Outcome is based on the Per-Protocol-Population (all randomized subjects without major protocol deviation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 1 x 12 mcg | IC51 2x6 mcg | IC51 1x6 mcg
Number analyzed (Participants) | 115 | 115 | 119
percentage of participants | 41.2 [32.2 to 50.3] | 97.3 [94.4 to 100.0] | 25.6 [17.7 to 33.6]
Statistical Analysis 1: Comparison: IC51 1 x 12 mcg vs IC51 2x6 mcg; Test type: Non-Inferiority or Equivalence — Assessment of non-inferiority of IC51 1x12 mcg vs. IC51 2x6 mcg at Day 56 based on the difference (IC51 1x12 mcg - IC51 2x6 mcg) in SCRs in the PP population. Non-inferiority of IC51 1 x 12 mcg compared to IC51 2 x 6 mcg was accepted if the lower limit of the 95% CI of the adjusted for center SCR difference (IC51 1 x 12 mcg - IC51 2 x 6 mcg) was higher than the noninferiority margin at -10%; p > 0.99, Mantel Haenszel

2. Secondary Outcome: SCR at Day 10, 28 and 35
Time Frame: Day 10, 28 and 35
Reporting Status: Not Posted

3. Secondary Outcome: GMT at Day 10, 28, 35 and 56
Time Frame: Day 10, 28, 35 and 56
Reporting Status: Not Posted

4. Secondary Outcome: Safety
Description: AEs, Local and systemic tolerability, Safety laboratory parameters
Time Frame: Study duration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IC51 2 x 6 mcg | IC51 1 x 12 mcg | IC51 1 x 6 mcg
Serious Adverse Events (participants affected / at risk) | 0/125 | 1/125 | 0/124
Other Adverse Events (participants affected / at risk) | 78/125 | 82/125 | 78/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 2 x 6 mcg (N=125) | IC51 1 x 12 mcg (N=125) | IC51 1 x 6 mcg (N=124)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 2 x 6 mcg (N=125) | IC51 1 x 12 mcg (N=125) | IC51 1 x 6 mcg (N=124)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (26) | 37 (41) | 36 (40)
Influenza like illness (General disorders) | 21 (22) | 27 (31) | 22 (26)
Fatique (General disorders) | 9 (12) | 18 (21) | 11 (11)
Headache (Nervous system disorders) | 30 (40) | 34 (49) | 34 (51)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other